CLINICAL TRIAL: NCT02917928
Title: The Potential of Carnosine Supplementation in Optimising Cardiometabolic Health in Patients With Prediabetes and Type 2 Diabetes: a Randomsied, Double-blinded, Placebo-controlled Trial
Brief Title: The Potential of Carnosine Supplementation in Optimising Cardiometabolic Health
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Monash University (Other)
Responsible Party: Principal Investigator, Barbora de Courten, Professor, Monash University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16061AI
Record Dates: First submitted 2016-09-19; First posted 2016-09-28 (Estimated); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Poor Glycemic Control; Cardiovascular Risk Factors; Cognitive Function 1, Social
Keywords: carnosine, type 2 diabetes, cardiovascular factors
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Carnosine; Methylcellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Active Comparator): Each participant will be given a daily oral dose 2 g of carnosine (4 tablets of 500mg each) for 14 weeks
  Interventions: Dietary Supplement: carnosine
- Control (Placebo Comparator): Each participant will be given a daily oral dose 2 g of placebo (4 tablets of 500mg each) for 14 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: carnosine — Each participant will be given a daily oral dose 2 g of carnosine (4 tablets of 500mg each) for 14 weeks
  Other Names: Pure Carnosine
  Arms: Intervention
Drug: Placebo — Each participant will be given a daily oral dose 2 g of placebo (4 tablets of 500mg each) for 14 weeks
  Other Names: Methylcellulose
  Arms: Control

SUMMARY:
The investigators hypothesise that carnosine supplementation will improve:

1. glycaemic control
2. cardiovascular risk factors
3. cognitive outcomes

in patients with prediabetes and type 2 diabetes, and this will be modulated by reduction in chronic low grade inflammation, oxidative stress and circulating advanced glycation end products levels.

3. Aims

To determine the potential of carnosine supplementation for 14 weeks to improve glycaemic control in type 2 diabetes, reduce risk factors for cardiovascular disease and improve cognitive function as well as identify metabolic pathways involved, specifically by:

1. Improving glycaemic control (HBA1c, fasting and 2 hour glucose and glucose area under the curve after oral glucose tolerance test)
2. Reducing cardiovascular risk factors (lipids; arterial (aortic) stiffness; central blood pressure (cBP); endothelial function).
3. Improve cognitive function (global cognitive score formed by a composite of 4 cognitive tests)
4. Decrease the chronic low grade inflammation, oxidative stress, advanced glycation end products, and advanced lipoxidation end products, and increase detoxification of reactive carbonyl species (RCSs).

DETAILED DESCRIPTION:
Type 2 diabetes is a major public health problem worldwide. Obesity itself markedly increases the risk of type 2 diabetes (DM2), which now affects every second obese person. With 60% of adult Australians overweight or obese and 25% of Australians aged over 25 years having prediabetes or diabetes, the quality-of-life and cost impact is inescapable. In Australia, direct healthcare costs for DM2 are currently estimated as $1.1 billion annually, with the prospect of doubling by 2025. Obesity and DM2 dramatically increase the risk of cardiovascular disease (CVD) with ~80% of individuals with both obesity and DM2 develop CVD. The annual healthcare costs for CVD in Australia now amount to $7.7 billion; and the total aggregated costs, including loss of income, are much higher again. Treating DM2 and CVD is expensive and often unsatisfactory. Weight loss and exercise are the mainstay of prevention and therapy but they are difficult and costly to achieve on a large scale; hence the DM2 epidemic continues unabated. Therefore, interventions at low cost and easy to implement at the population level is urgently required.

Neurodegenerative diseases often occurs in people with DM2, and DM2 is in turn associated with increased risk of cognitive decline. Neurodegenerative diseases such as Alzheimer's disease are also associated with metabolic impairment. They share many common pathogenic features with DM2 such as insulin resistance, chronic low-grade inflammation, vascular disease, oxidative stress and accumulation of advanced glycation endproducts (AGEs). Progression of these diseases over years-decades is also worsened by a sedentary life-style. Therefore not surprisingly, regular physical activity is beneficial in those patients, likely due to improvement of neurological, motor and cardiometabolic profile. However, it is difficult and costly to achieve on a large scale, and thus, safe and low-cost strategies are needed.

Type 2 diabetes is associated with increased amounts of ectopic fat depots in muscle including intramyocellular lipids (IMCL), and adipocytes located between muscle groups (inter-muscular) and also between muscle fascicles (intramuscular). Both IMCL and intra- and inter-muscular adipose tissue (IMAT) may deleteriously effect muscle metabolism and insulin sensitivity through increased local secretion of pro-inflammatory adipokines, and inter-muscular fat may additionally impair insulin action through reductions in blood flow to muscle.

Could carnosine be that strategy? Strong molecular and animal data (>2000 papers) suggests that it has great potential, with all the relevant properties. Carnosine, is present in several tissues including muscle and brain, easily crosses the blood-brain barrier, and extensive animal data show that carnosine has chelating properties and modulates glucose metabolism, advanced glycation, pro-inflammatory and pro-oxidative states, as well as motor functions and neurotransmission. A promising further use may derive from its effect on cardiometabolic health and neuroprotection. Current research, confined to animal studies, supports carnosine supple¬ment¬ation for preventing and treating obesity, DM2, CVD, and neurodegenerative diseases - by virtue of its anti-inflammatory, antioxidative, anti-glycating and chelating effects. Our team's novel pilot studies provide the first human cross-sectional and interventional metabolic data, and demonstrate relationships among carnosine, obesity, insulin resistance, and dyslipidaemia. Previous clinical trials also showed that supplementation of carnosine for 2-3 months improved cognitive performance in healthy individuals and patients with neurodegenerative diseases. However, none of them showed its effect in patient with type 2 diabetes and explored the effects of change in cardiometabolic outcomes on cognitive function.

Apart from its excellent side-effect profile, carnosine is cheap and safe (it is an over-the-counter dietary supplement), making it prima facie ideal for widespread, low cost use. Robust human research is now urgently needed to test the therapeutic potential of carnosine in improving cardiometabolic profile and cognitive function, and study the mechanisms involved.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 or <=70 years
* Weight change < 5 kg in last 6 months
* HbA1c level <= 8%
* Patients with prediabetes (Impaired glucose tolerance and impaired fasting glycaemia) or type 2 diabetes (diet controlled or on oral therapy)
* Patients will have to be on oral therapy for diabetes (without changes in treatment) at least for 3 months.
* Patients will be advised not to change their pre-existing therapy for diabetes and cardiovascular risk factors for the duration of the study if HbA1c is not above 8%
* No recent blood transfusion (3 months)
* No current intake of anti-inflammatory medications and supplements
* No significant kidney, cardiovascular, haematological, respiratory, gastrointestinal, or central nervous system disease, as well as no psychiatric disorders, no active cancer within the last five years; no presence of acute inflammation (by history, physical or laboratory examination)
* Pregnant or lactating

Exclusion Criteria:

* Age <18 or > 70 years
* HbA1c level of >= 8%
* Weight change > 5 kg in last 6 months
* Morbid obesity (body mass index >40 kg/m2)
* Current smoking habit and high alcohol use
* Patients on insulin
* Taking anti-inflammatory medications or supplements
* Recent blood transfusion history
* Kidney (estimated glomerular filtration rate < 30 ml/min), cardiovascular, haematological, respiratory, gastrointestinal, or central nervous system disease, as well as psychiatric disorder, active cancer within the last five years; presence of acute inflammation (by history, physical or laboratory examination)
* Pregnancy or lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-10; Primary Completion 2023-01 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Change in Oral Glucose Tolerance Test | baseline and 14 weeks
  After a 10-12 h overnight fast, participants will ingest 75g of glucose over 2 mins. Blood samples will be drawn at 0, 30, 60, 90 and 120 min for plasma glucose and insulin concentrations. We will evaluate the area under the curve.

SECONDARY OUTCOMES:
Change in HbA1c | baseline and 14 weeks
  Blood samples will be measured using High Performance Liquid Chromatography.
Change in lipid profile | baseline and 14 weeks
  Blood samples will be analysed using High Performance Liquid Chromatography
Change in systolic and diastolic blood pressure | baseline and 14 weeks
  Resting systolic and diastolic blood pressure and pulse rate will be measured using an automated oscillometric measurement system (Dinamap, USA) after a 30 minute rest.
Change in arterial stiffness and central blood pressure | baseline and 14 weeks
  Aortic (carotid-femoral) pulse wave velocity (aPWV) will be measured using the non-invasive Complior device (Alam Medical, French).
Change in markers of endothelial dysfunction | baseline and 14 weeks
  This is done using non-invasive peripheral arterial tomography (PAT; endothelium-dependent digital pulse amplitude testing (EndoPAT), Itamar Medical Ltd, Israel), which records continuous plethysmographic signals of the finger arterial pulse wave. Finger plethysmographic probes are placed on each index finger; and after a 5 min equilibration period, a blood pressure cuff on the non-dominant arm is inflated to 60 mmHg above systolic for 5 min and then deflated to induce reactive hyperaemia. Measurements of post-occlusion changes (reactive hyperaemia PAT: RH-PAT) are continued for 10 min. Results are normalised to the non-occluded arm, compensating for potential systemic changes (RH-PAT ratio).
Change in heart rate variability | baseline and 14 weeks
  The Zephyr Biomodule BH3 (Black Sensor, produced by Zephyr Technology) will be used to measure heart rate and heart rate variability for three consecutive days.
Change in interleukins | baseline and 14 weeks
  Interleukins will be measured by quantitative sandwich enzyme immunoassays (R & D Systems Inc, USA).
Change in tumour necrosis factor α | baseline and 14 weeks
  Tumour necrosis factor α (TNFα) will be measured by quantitative sandwich enzyme immunoassays (R & D Systems Inc, USA).
Change in macrophage migration inhibitory factor | baseline and 14 weeks
  Macrophage migration inhibitory factor will be measured by quantitative sandwich enzyme immunoassays (R & D Systems Inc, USA).
Change in plasma C- reactive protein | baseline and 14 weeks
  Plasma C- reactive protein (hsCRP) will be measured using high sensitivity assay (BN-II nephelometer; Dade Behring Diagnostics, NSW).
Change in plasma and urinary advanced glycation end products | baseline and 14 weeks
  Measured by liquid chromatography-tandem mass spectrometry and ELISA tests. Circulating receptor for AGEs will be measured by ELISA. Protein modifications and the effect of carnosine supplementation will be determined by proteomic approaches.
Change in plasma and urinary advanced lipoxidation end products | baseline and 14 weeks
  This will be determined by measuring the advanced oxidation protein products and by measuring the cysteinate form of albumin by mass spectrometry. Mercapturic acid adducts with the main reactive carbonyls species will also be quantitatively determined by liquid chromatography electrospray ionization mass spectrometry/mass spectrometry analysis (LC-MS/MS).
Change in general cognitive function | baseline and 14 weeks
  Participants' cognitive function will be assessed using Cambridge Neuropsychological Test Automated Battery (CANTAB) battery for Prodromal Alzheimer's disease, Victoria Stroop test, Trail Making Test and Digit Symbol Substitution Test.

OTHER OUTCOMES:
Change in liver stiffness and fat | baseline and 14 weeks
  A non-invasive transient elastography (Fibroscan, EchoSens, Paris) will be used to assess liver fibrosis based on the measurement of liver fat and stiffness
Change in Serum and urine carnosine | baseline and 14 weeks
  This will be measured by ELISA for human carnosinase 1 (CN1) with a monoclonal antibody (clone ATLAS, Abcam plc) and peroxidase substrate .
Change in skeletal muscle fat and density | baseline and 14 weeks
  We will also measure the change in muscle and fat tissue density of participants' non-dominant leg using Quantitative Computed Tomography (pQCT). Participants will be seated in their non-dominant leg positioned inside the machine gantry. Muscle cross sectional area (mm2) and muscle density (mg/cm3) will be determined using the manufacturer's algorithms.
Change in body composition | baseline and 14 weeks
  body composition by dual energy x-ray absorptiometry (DEXA), which is a non-invasive assessment of soft tissue composition by region with a precision of 4-5%; central adiposity assessed in duplicate using a constant-tension tape for taking waist, and hip circumference. Bioimpedance measurement will be also collected for validation purposes.

CONTACTS AND LOCATIONS:
Overall Officials: Barbora de courten, MD,PHD,MPH, Principal Investigator — Monash University
Locations (1):
- Monash Centre for Health Research and Implementation, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saadati S, Jansons P, Scott D, de Courten M, Mousa A, Feehan J, Mesinovic J, de Courten B. The Effect of Carnosine Supplementation on Musculoskeletal Health in Adults with Prediabetes and Type 2 Diabetes: A Secondary Analysis of a Randomized Controlled Trial. Nutrients. 2024 Dec 15;16(24):4328. doi: 10.3390/nu16244328. PMID 39770949
- [Derived] Saadati S, de Courten M, Deceneux C, Plebanski M, Scott D, Mesinovic J, Jansons P, Aldini G, Cameron J, Feehan J, Mousa A, de Courten B. Carnosine Supplementation Has No Effect on Inflammatory Markers in Adults with Prediabetes and Type 2 Diabetes: A Randomised Controlled Trial. Nutrients. 2024 Nov 15;16(22):3900. doi: 10.3390/nu16223900. PMID 39599686
- [Derived] Saadati S, Cameron J, Menon K, Hodge A, Lu ZX, de Courten M, Feehan J, de Courten B. Carnosine Did Not Affect Vascular and Metabolic Outcomes in Patients with Prediabetes and Type 2 Diabetes: A 14-Week Randomized Controlled Trial. Nutrients. 2023 Nov 19;15(22):4835. doi: 10.3390/nu15224835. PMID 38004228
- [Derived] Baye E, Menon K, de Courten MP, Earnest A, Cameron J, de Courten B. Does supplementation with carnosine improve cardiometabolic health and cognitive function in patients with pre-diabetes and type 2 diabetes? study protocol for a randomised, double-blind, placebo-controlled trial. BMJ Open. 2017 Sep 1;7(9):e017691. doi: 10.1136/bmjopen-2017-017691. PMID 28864708